CLINICAL TRIAL: NCT00969540
Title: Double Blind, Placebo Controlled, Crossover Pilot Trial on the Effect of Optically Modified Polyethylene Terephthalate Fiber Mattress Covers on Sleep Disturbances in Patients With Chronic Back Pain
Brief Title: Trial on the Effect of Optically Modified Fiber Mattress Covers on Sleep Disturbances in Patients With Chronic Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Annabel Kim Wang, Associate Clinical Professor, University of California, Irvine
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: mattress1
Record Dates: First submitted 2009-08-31; First posted 2009-09-01 (Estimated); Results first posted 2014-12-03 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Back Pain; Insomnia
Keywords: Back Pain; Sleep
MeSH Terms: conditions — Back Pain; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Mattress Cover (Active Comparator): Subjects in this arm will be given the placebo mattress cover followed active mattress cover .
  Interventions: Device: Active Mattress Cover
- Placebo Mattress Cover (Placebo Comparator): Subjects in this arm will be given the active mattress cover followed by the placebo mattress cover.
  Interventions: Device: Placebo Mattress Cover

INTERVENTIONS:
Device: Active Mattress Cover — Active Mattress Cover
  Arms: Active Mattress Cover
Device: Placebo Mattress Cover — Placebo Mattress Cover
  Arms: Placebo Mattress Cover

SUMMARY:
Sleep quantity and quality can be influenced by the type of mattress used. This study is being done to see if a mattress cover with optically active particles can help back pain and improve sleep quality.

DETAILED DESCRIPTION:
It is commonly observed that sleep in its quantity and quality is influenced by the type of mattress used at night. A recent study in patients with back pain showed that waterbeds and foam mattresses did influence back symptoms, function and sleep more positively than did a hard mattress. Pain improves with airbeds compared to regular innerspring mattresses. This study will analyze the effect of optically active particles mattress covers on sleep. The researcher is interested in learning if regular mattress or the study mattress cover (containing optically modified polyethylene terephthalate fiber mattress cover) is more useful in helping back pain and sleep quality.

ELIGIBILITY:
Inclusion Criteria:

You are eligible to participate in this study if you:

1. have a clinical diagnosis of chronic lower back pain
2. have pain measured on the Visual Analogue scale
3. have sleep disturbances at night associated with chronic lower back pain
4. are 18 years or older
5. sign the written, informed consent form prior to the initiation of any study procedures
6. have an habitual bedtime between 8 P.M. and 12 A.M.
7. are on a stable pain management regime

Exclusion Criteria:

You are not eligible to participate in this study if you:

1. are unwilling or unable to comply with the protocol or scheduled appointments
2. are unable to understand the language in which the approved informed consent is written
3. have no pain measured on the Visual Analogue scale
4. are unable to walk, wheel chair bound or confined to bed
5. are deemed by the investigator to be unreliable to wear the actigraphy, to complete the sleep log, to use the provided mattress covers at the proper time, to come to the scheduled visits or to answer questions regarding the subject's condition or medication use
6. lack a mobile arm to which to attach an actigraphy.
7. are currently participate or participated in another clinical study within the past 30 days
8. demonstrate an unwillingness to comply with the maximum limit of two alcoholic drinks per day and only 1 alcoholic drink after 6:00 P.M. for the duration of the protocol
9. use tobacco products or any other products during nightly awakenings that may interfere with the sleep wake cycle
10. have any unstable medical condition as determined by the investigator, or any other serious disease or condition that might affect life expectancy or make it difficult to successfully manage and follow the subject according to the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annabel K Wang, MD, Principal Investigator — UC Irvine
Locations (1):
- UC Irvine-MDA ALS and Neuromuscular Center, Orange, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was by advertisement.
Pre-assignment Details: A total of 8 participants were entered into this crossover study. The total duration of the study was approximately 49 days, including 14 days of screening and 14 days of the first intervention, 7 days of washout, and 14 days of the second intervention.
Groups:
- Placebo Mattress Cover First, Then Active Mattress Cover: Subjects were randomly assigned in this crossover double blind designed trial to the placebo mattress cover or active mattress cover for 14 days.
- Active Mattress Cover First, Then Placebo Mattress Cover: Subjects were randomly assigned in this crossover double blind designed trial to the active mattress cover or placebo mattress cover for 14 days.
Period: Overall Study
Arm/Group | Placebo Mattress Cover First, Then Active Mattress Cover | Active Mattress Cover First, Then Placebo Mattress Cover
Started | 4 | 4
Completed | 3 | 3
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo Mattress Cover First, Then Active Mattress Cover: Subjects in this crossover double blind designed trial will be randomized into the placebo mattress cover group for 14 days. After a 7 day washout, they will be entered into the active mattress cover group for 14 days.
- Active Mattress Cover First, Then Placebo Mattress Cover: Subjects in this crossover double blind designed trial will be randomized into the active mattress cover group for 14 days. After a 7 day washout, they will be entered into the placebo mattress cover group for 14 days.
- Total: Total of all reporting groups
Arm/Group | Placebo Mattress Cover First, Then Active Mattress Cover | Active Mattress Cover First, Then Placebo Mattress Cover | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (13) | 48 (7) | 47 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Optically Modified Polyethylene Terephthalate Fiber Mattress Cover (OMPETFMC) Improves Sleep Quality in Patients With Lower Back Pain as Measured by Clinical Global Impression (CGI).
Description: The primary outcomes are the change in mean daily Clinical Global Impressions (pain and sleep) in placebo mattress compared to active mattress cover (assessed daily for 14 days per intervention).
  The daily scores range from 1 (very much improved) to 7 (very much worse).
Time Frame: 14 days
Population: The sponsor determined the size of the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Mean CGI Pain Scores With Placebo Mattress Cover.: Mean Clinical Global Impression pain scores with placebo mattress cover.
- Mean CGI Pain Scores With Active Mattress Cover.: Mean Clinical Global Impression pain scores with active mattress cover.
- Mean CGI Sleep Scores With Placebo Mattress Cover.: Mean Clinical Global Impression sleep scores with placebo mattress cover.
- Mean CGI Sleep Scores With Active Mattress Cover.: Mean Clinical Global Impression sleep scores with active mattress cover.
Arm/Group | Mean CGI Pain Scores With Placebo Mattress Cover. | Mean CGI Pain Scores With Active Mattress Cover. | Mean CGI Sleep Scores With Placebo Mattress Cover. | Mean CGI Sleep Scores With Active Mattress Cover.
Number analyzed (Participants) | 6 | 6 | 6 | 6
units on a scale
  Subject 1 | 4.07 (1.27) | 3.86 (1.10) | 3.93 (1.27) | 3.86 (1.10)
  Subject 2 | 3.86 (0.53) | 3.86 (0.66) | 3.86 (0.77) | 3.93 (0.62)
  Subject 3 | 4.00 (0.00) | 4.00 (0.00) | 3.92 (0.29) | 4.00 (0.00)
  Subject 4 | 4.00 (0.00) | 4.07 (0.27) | 4.00 (0.00) | 4.00 (0.00)
  Subject 5 | 3.00 (0.00) | 3.00 (0.00) | 3.14 (0.53) | 3.00 (0.00)
  Subject 6 | 4.00 (0.00) | 4.00 (0.00) | 4.00 (0.00) | 4.00 (0.00)

2. Secondary Outcome: Sleep Variables (Nighttime Wake-time) Measured With Actigraphy in Patients With Lower Back Pain.
Description: Secondary outcome: Nighttime wake-time after sleep onset with placebo mattress cover compared to active mattress cover.
Time Frame: Assessed daily for 14 days per intervention.
Population: The sponsor determined the number of participants.
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- Nighttime Wake Time With Placebo Mattress Cover: Nighttime wake time after sleep onset with placebo mattress cover.
- Nighttime Wake Time With Active Mattress Cover: Nighttime wake time after sleep onset with active mattress cover.
Arm/Group | Nighttime Wake Time With Placebo Mattress Cover | Nighttime Wake Time With Active Mattress Cover
Number analyzed (Participants) | 6 | 6
Minutes
  Subject 1 | 53.38 (26.70) | 71.31 (28.42)
  Subject 2 | 59.15 (19.72) | 107.38 (50.76)
  Subject 3 | 113.83 (34.37) | 128.38 (77.08)
  Subject 4 | 50.23 (35.30) | 76.09 (37.27)
  Subject 5 | 44.91 (50.58) | 49.92 (38.70)
  Subject 6 | 71.75 (25.11) | 80.58 (27.49)

3. Secondary Outcome: Sleep Variables (Total Sleep) Measured With Actigraphy in Patients With Lower Back Pain.
Description: Secondary outcome: Total sleep time with placebo mattress cover compared to active mattress cover.
Time Frame: Assessed daily for 14 days per intervention.
Population: The sponsor determined the number of participants.
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- Total Sleep With Placebo Mattress Cover: Total sleep with placebo mattress cover (minutes).
- Total Sleep With Active Mattress Cover: Total sleep with active mattress cover (minutes).
Arm/Group | Total Sleep With Placebo Mattress Cover | Total Sleep With Active Mattress Cover
Number analyzed (Participants) | 6 | 6
Minutes
  Subject 1 | 433.15 (110.80) | 435.92 (75.93)
  Subject 2 | 406.54 (46.23) | 384.00 (113.18)
  Subject 3 | 447.83 (190.13) | 435.46 (103.15)
  Subject 4 | 401.54 (61.69) | 400.73 (45.71)
  Subject 5 | 476.45 (87.86) | 451.85 (95.54)
  Subject 6 | 394.67 (94.64) | 341.75 (71.75)

4. Secondary Outcome: Sleep Variables (Nocturnal Awakenings) Measured With Actigraphy in Patients With Lower Back Pain.
Description: Secondary outcome: Number of nocturnal awakenings with placebo mattress cover compared to active mattress cover.
Time Frame: Assessed daily for 14 days per intervention.
Population: The sponsor determined the number of participants.
Measure: Mean (Standard Deviation); unit: Awakenings
Groups:
- Nocturnal Awakenings With Placebo Mattress Cover: Number of nocturnal awakenings with placebo mattress cover.
- Nocturnal Awakenings With Active Mattress Cover: Number of nocturnal awakenings with active mattress cover.
Arm/Group | Nocturnal Awakenings With Placebo Mattress Cover | Nocturnal Awakenings With Active Mattress Cover
Number analyzed (Participants) | 6 | 6
Awakenings
  Subject 1 | 19.85 (10.53) | 23.46 (8.36)
  Subject 2 | 10.62 (2.40) | 12.31 (4.13)
  Subject 3 | 19.08 (5.32) | 22.23 (11.06)
  Subject 4 | 20.38 (12.59) | 26.27 (9.88)
  Subject 5 | 10.73 (10.14) | 10.54 (7.49)
  Subject 6 | 17.17 (4.84) | 18.25 (6.33)

5. Secondary Outcome: Sleep Variables (Sleep Efficiency) Measured With Actigraphy in Patients With Lower Back Pain.
Description: Secondary outcome: Sleep efficiency in placebo mattress cover compared to active mattress cover.
Time Frame: Assessed daily for 14 days per intervention.
Population: The sponsor determined the number of participants.
Measure: Mean (Standard Deviation); unit: Percentage of time asleep
Groups:
- Sleep Efficiency With Placebo Mattress Cover: Sleep efficiency with placebo mattress cover.
- Sleep Efficiency With Active Mattress Cover: Sleep efficiency with active mattress cover.
Arm/Group | Sleep Efficiency With Placebo Mattress Cover | Sleep Efficiency With Active Mattress Cover
Number analyzed (Participants) | 6 | 6
Percentage of time asleep
  Subject 1 | 88.17 (5.51) | 85.65 (5.62)
  Subject 2 | 87.28 (2.76) | 76.72 (14.18)
  Subject 3 | 79.35 (9.30) | 75.95 (14.84)
  Subject 4 | 88.37 (7.64) | 84.00 (7.68)
  Subject 5 | 90.85 (10.28) | 89.58 (8.28)
  Subject 6 | 83.79 (2.53) | 79.67 (6.02)

6. Secondary Outcome: Sleep Variables (Sleep Latency) Measured With Actigraphy in Patients With Lower Back Pain.
Description: Secondary outcome: Sleep latency in placebo mattress cover compared to active mattress cover.
Time Frame: Assessed daily for 14 days per intervention.
Population: The sponsor determined the number of participants.
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- Sleep Latency With Placebo Mattress Cover: Sleep latency with placebo mattress cover (minutes).
- Sleep Latency With Active Mattress Cover: Sleep latency with active mattress cover (minutes).
Arm/Group | Sleep Latency With Placebo Mattress Cover | Sleep Latency With Active Mattress Cover
Number analyzed (Participants) | 6 | 6
Minutes
  Subject 1 | 2.92 (5.06) | 1.46 (2.50)
  Subject 2 | 1.15 (3.36) | 0 (0)
  Subject 3 | 9.75 (18.86) | 7.54 (18.33)
  Subject 4 | 2.69 (9.71) | .27 (0.90)
  Subject 5 | 0.91 (2.43) | 0.15 (0.55)
  Subject 6 | 4.83 (7.03) | 5.17 (10.66)

ADVERSE EVENTS:
Time Frame: 1 year 2 months (April 2010-June 2011)
Groups:
- Placebo Mattress Cover: Subjects will be randomly assigned in this crossover double blind designed trial to the placebo mattress cover for 14 days, followed by the active mattress cover for 14 days after a 7 day wash out period.
- Active Mattress Cover: Subjects will be randomly assigned in this crossover double blind designed trial to the active mattress cover for 14 days, followed by the placebo mattress cover for 14 days after a 7 day wash out period.
Arm/Group | Placebo Mattress Cover | Active Mattress Cover
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3

LIMITATIONS AND CAVEATS:
This is a pilot study to determine the framework to study sleep, pain and mattress covers. The number of subjects is small. The observed data is evaluated in a descriptive (bar graph) presentation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other